CLINICAL TRIAL: NCT01355978
Title: Acceptability, Comfort, and Exercise Tolerance Using a Non-invasive Ventilation System in Patients With Moderate-to-Severe COPD (PRIDE)
Brief Title: Non-invasive Ventilation System in Moderate-to-Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breathe Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP-00-0031
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Airflow Obstruction, Chronic; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noninvasive Open Ventilation System (Experimental): Portable noninvasive open ventilator & nasal interface.
  Interventions: Device: Noninvasive Open Ventilation System

INTERVENTIONS:
Device: Noninvasive Open Ventilation System — Noninvasive ventilation system

SUMMARY:
When using the Breathe Technologies Ventilation System during simulated activities of daily living (ADLs), Subjects with moderate-to-severe chronic obstructive pulmonary Disease (COPD) will be comfortable and report acceptability.

DETAILED DESCRIPTION:
The primary objective of the study was to evaluate the Breathe Technologies Ventilator System with regard to subject acceptability, comfort, and effect on exercise and activities of daily living tolerance.

Primary Hypothesis:

1. When using the Breathe Technologies Ventilation System during simulated activities of daily living (ADL), Subjects with moderate-to-severe COPD will be comfortable and report acceptability.

   Secondary Hypotheses:
2. When using the Breathe Technologies Ventilation System during simulated ADLs, Subjects with moderate-to-severe COPD will experience tolerable dyspnea as measured using the Borg Dyspnea Score (BDS) and a visual analog Comfort Scale (VACS).
3. Subjects will prefer using the Breathe Technologies Ventilation System over standard oxygen therapy during exertion and during ADLs after using the ventilator therapy for five days.

ELIGIBILITY:
Inclusion Criteria:

* Have participated and completed the NOVEL 1 or NOVEL 2 studies.
* Be 21-80 years of age (inclusive) at time of informed consent.
* Require nasal oxygen of ≥ 2 LPM during exertion, and ≥ 1 LPM at rest.
* Exhibit dyspnea and have lung disease process dominated by COPD per the Study Investigator.
* Have a self-reported MMRC Dyspnea Score ≥ 2 on a scale of 0-4.
* Have spirometric evidence of COPD with an FEV1 of < 50% predicted and FEV1/FVC < 0.70, measured within the last 6 months (GOLD stage III and IV).
* Have a resting respiratory rate of less than or equal to 30 bpm.
* Be fluent in reading and speaking the English language.
* Be able to clearly communicate and to indicate a self-assessment of dyspnea and/or fatigue.
* Be willing and able to participate in, and to complete all required study procedures, including the ability to pull an E-sized oxygen cylinder.
* Report having a smoking history of ≥ 10 pack-years.
* Provide written informed consent to participate in the study.

Exclusion Criteria:

Subject must NOT meet any of the following criteria, or they will be excluded from study participation:

* Be a current tobacco smoker
* Have a history of pneumothorax in last 2 years.
* Have a history of severe, giant bullae.
* Have a history of unstable angina
* Reports the onset of cardiac arrhythmia(s) within the past 7 days.
* Report having serious epistaxis within the last 10 days.
* Have a history of severe pulmonary hypertension and/or NYHA Stage III and IV decompensated heart failure.
* Reports symptoms of acute COPD exacerbation within the past 48 hours.
* Have been discharged from the hospital within 30 days of screening for infection or acute illness or COPD exacerbation.
* Have a prescription or history of requiring > 8 LPM oxygen during exertion.
* Have a history of serious allergic airways disease (e.g., high eosinophil count or elevated IgE).
* Report or have evidence of LVEF < 30 %
* Have a BMI > 40
* Have a history of thoracotomy, sternotomy, major cardiopulmonary intervention (e.g., lung resection, open heart surgery), or any procedure 6 months before study entry likely to cause instability of pulmonary status.
* Have a history of lung disease unrelated to smoking that affects oxygenation or survival.
* Is participating in another intervention study or have participated within 90 days of enrollment.
* Have endobronchial valves or other bronchial tree implants such as stents.
* Have a disease or condition expected to cause death, inability to perform procedures for the trial, or inability to comply with the therapy.
* Have a history of intolerance to oxygen therapy.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kops, MD, Principal Investigator — John Muir Health; Lynn McCabe, RRT, RCP, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - John Muir Health, Concord, California
  - Sharp Memorial Hospital, San Diego, California
  - McKay-Dee Hospital Center, Ogden, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Noninvasive Open Ventilation System
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Adult subjects with chronic obstructive lung disease.
Groups:
- Noninvasive Open Ventilation System: Portable noninvasive open ventilator & nasal interface. Noninvasive Open Ventilation System used during activities of daily living.
Arm/Group | Noninvasive Open Ventilation System
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Device Tidal Volume
Description: Evaluate the mean test volume for three activity levels. Subjects completed five consecutive, 6-hour clinic days in which the NIOV system was worn continuously while at rest, during activities of daily living (ADLs).
Time Frame: Periodically over six hours x 5 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Noninvasive Open Ventilation System
Number analyzed (Participants) | 18
mL | 180 (24)

2. Secondary Outcome: Device Preference
Description: 5-point Likert Scale completed at the end or the 5-day study period
  - Preference Scale: 5 = Max preference (Prefer to use the test device), 1 = Min preference (Do not prefer to use the test device)
Time Frame: At conclusion of subject's participation (up to two weeks)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Noninvasive Open Ventilation System
Number analyzed (Participants) | 18
units on a scale | 4 [3 to 5]

3. Secondary Outcome: Safety and Device-related Adverse Events
Description: Any adverse events reported during he study period.
Time Frame: Continuous from Study Day 2 through Study Day 6
Measure: Number; unit: participants
Arm/Group | Noninvasive Open Ventilation System
Number analyzed (Participants) | 18
participants | 3

ADVERSE EVENTS:
Time Frame: Continuously for 1 week, starting a screening visit through end of study (Day 6).
Arm/Group | Noninvasive Open Ventilation System
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Noninvasive Open Ventilation System (N=18)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — For Subject JM003, a mild skin rash was noted on the finger on which the pulse oximeter probe was attached. The probe was relocated and the rash resolved without intervention.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (18) — Subject SH011 reported being SOB following exercising on treadmill. SOB resolved after discontinuing exercise. No intervention was required.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (18) — Subject JM008 reported being SOB during performance of simulated activity of daily living (vacuuming). SOB resolved quickly when ADL was stopped. No other intervention was required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No